CLINICAL TRIAL: NCT02366156
Title: A Randomized, Double-Blind, 3-Period Crossover Study to Evaluate the Effects of a Dietary Supplement Containing Botanical Extracts on Fasting and Postprandial Lipid Metabolism in Apparently Healthy, Overweight and Obese Individuals
Brief Title: A 12 Week, 3-Period Study to Evaluate the Effects of a Dietary Supplement on Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BIO-1403
Record Dates: First submitted 2014-10-15; First posted 2015-02-19 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Inactive capsules
  Interventions: Dietary Supplement: Placebo
- Low Dose Grape Blend (Active Comparator): Low dose grape blend providing 375 mg whole grape extract + 375 mg grape seed extract/d (750 mg total botanical extracts/d).
  Interventions: Dietary Supplement: Low Dose Grape Blend
- High Dose Grape Blend (Active Comparator): High dose grape blend providing 500 mg whole grape extract + 500 mg grape seed extract/d (1000 mg total botanical extracts/d)
  Interventions: Dietary Supplement: High Dose Grape Blend

INTERVENTIONS:
Dietary Supplement: Placebo — Three placebo capsules consumed prior to breakfast each day for 4 weeks
  Arms: Placebo
Dietary Supplement: Low Dose Grape Blend — Three low dose grape blend capsules consumed prior to breakfast each day for 4 weeks.
  Arms: Low Dose Grape Blend
Dietary Supplement: High Dose Grape Blend — Three high dose grape blend capsules consumed prior to breakfast each day for 4 weeks.
  Arms: High Dose Grape Blend

SUMMARY:
This study will evaluate the effects of encapsulated botanical extracts, previously shown to inhibit the enzyme diacylglycerol-acyltransferase-1 (DGAT-1) in vitro, on fasting and postprandial lipid metabolism during an oral fat tolerance test (OFTT) in apparently healthy, overweight and obese adult men and women.

DETAILED DESCRIPTION:
Medications currently approved for the treatment of obesity act primarily to promote a state of energy balance - by either suppressing appetite or interfering with lipid absorption in the small intestine. Similarly, it may be possible to reduce or inhibit the synthesis of triglycerides (TG) from dietary fat by targeting the activity of diacylglycerol-acyltransferase-1 (DGAT-1) in the enterocytes of the small intestine.

DGAT-1 catalyzes the final step in the biosynthesis of TG and is most abundantly expressed in the small intestine and adipose tissue. DGAT-1 in enterocytes is critical for assembly of TG from fatty acids derived from food intake. Ingested dietary fat is cleaved to monoacylglycerol and free fatty acids by lipases in the gut lumen and these are next taken up by the enterocytes, where they are re-esterified to TG in the postprandial period. TG is eventually released into circulation, primarily transported by chylomicrons. Thus, DGAT-1 plays a critical role in the absorption of dietary fat and inhibition of DGAT-1 has been shown to delay and decrease re-esterification of dietary fats into circulating TG. It is hypothesized that this effect may lead to decreased deposition of excess dietary fat as adipose tissue, perhaps due to increased fatty acid oxidation in the enterocytes.

The potential physiological benefits of DGAT-1 inhibition lead to the development of the potent, selective DGAT-1 inhibitor, AZD7687. Human clinical trials of AZD7687 demonstrated attenuation of postprandial TG excursions, consistent with inhibition of gut DGAT-1. However, this compound has limited, if any, therapeutic potential due to profound gastrointestinal (GI) side effects, particularly diarrhea, nausea, and abdominal cramping which were deemed intolerable. Moreover, no consistent dose-related treatment effects on body weight, glucose or lipid metabolism were found in the small trials which were deemed to be non-representative of the target therapeutic population.

Both cell-free and cellular in vitro models have been used to identify botanical extracts that have potential to inhibit DGAT-1. In a follow-up 7-d parallel arm proof-of-mechanism human clinical trial, each of four lead ingredients (2 g/d) were evaluated for the ability to inhibit the intestinal release of dietary fat into circulation following a high-fat meal challenge using post-prandial TG response as a surrogate marker. Of the four lead botanical ingredients, whole grape extract (WGE) reduced fasting and postprandial TG levels (total area under the curve from 0 to 6 h) by ~ 7% to 8% following a high-fat meal challenge. This demonstration of efficacy, albeit modest, was sufficient to warrant continued exploration. Importantly, only a few subjects reported very mild GI side effects, primarily bloating, in this trial.

Combinations of WGE with other botanical extracts possessing biological activity against supportive secondary mechanisms that might strengthen the overall inhibition of dietary fat release into circulation and fat deposition were then explored. To examine potential synergistic interactions, WGE was combined with other ingredients known to act on complementary biological pathways that converge into a single efficacy outcome; in this case, cellular TG levels. Ingredients that had effects on both glucose and fatty acid metabolism that could ultimately synergize with the DGAT-1 pathway were chosen. The complementary pathway targets chosen for these experiments were Peroxisome-Proliferator-Activated Receptor-gamma Coactivator 1-alpha (PGC1-α) and Sterol Regulatory Element Binding Protein 1c (SREBP1c).

In the cellular DGAT-1 model, grape seed extract (GSE) resulted in a significant inhibition of DGAT-1 activity when combined with WGE. The combination index (CI), a quantitative measure of synergy, indicated a strong synergistic effect (CI = 0.61). Synergy occurred at a 1:1 ratio of WGE to GSE, and at ratios that induced no effect on DGAT-1 activity when either was used alone. The synergy data, together with the proof of mechanism clinical data, forms the basis for conducting the presently proposed clinical trial at a WGE level below that used in the previous study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18-70 years of age, inclusive.
2. Subject has a fasting TG concentration of ≥150 and <500 mg/dL at visit 1b (week -1). One venous retest allowed for 145-149 and 500-550 mg/dL values.
3. Subject has a body mass index (BMI) of 25.00-34.99 kg/m2 at visit 1b (week -1).
4. Subject is willing to maintain habitual diet and physical activity patterns during the study period.
5. Subject has no plans to change smoking habits during the study period, and if a current smoker, subject is willing to refrain from all tobacco products for 1 h prior to all clinic visits in addition to up to 9 h during the test visits.
6. Subject has a score of 7 to 10 on the Vein Access Scale at screening visit (visit 1b, week -1).
7. Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
8. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has abnormal laboratory test results of clinical significance at visit 1b (week -1), at the discretion of the Investigator. One re-test will be allowed on a separate day prior to visit 2 (week 0), for subjects with abnormal laboratory test results.
2. Subject has a history or presence of clinically important endocrine (including type 1 or 2 diabetes mellitus), cardiovascular (including, but not limited to history of myocardial infarction, peripheral arterial disease, stroke), pulmonary (including uncontrolled asthma), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric or biliary disorders.
3. Subject has a history or current GI disorder that, in the judgment of the Investigator, may have the potential to disrupt normal digestion and absorption of dietary fats, including, but not limited to, Crohn's disease, inflammatory bowel disease, irritable bowel syndrome, significant lactose intolerance and/or egg allergy.
4. Subject has a known genetic predisposition to hyperlipidemia - as diagnosed by a health care professional.

   Subject is a heavy smoker, defined as a history of smoking >1 pack-per-day in the 3 months prior to visit 1b (week -1).
5. Subject has a history of difficulty swallowing tablets/capsules that could affect ability to consume the study product.Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
6. Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian), in the opinion of the Investigator.
7. Subject has had a weight loss or gain >4.5 kg in the 3 months prior to visit 1b (week -1).
8. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at visit 1b (week -1). One re-test will be allowed on a separate day prior to visit 2 (week 0), for subjects whose blood pressure exceeds either of these cut points, in the judgment of the Investigator.
9. Subject has not been on a stable dose of antihypertensive medication (at least 4 weeks prior to visit 1b, week -1 and for the duration of the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Fasting triglycerides | Baseline and at the end of each 4 week treatment period for a total of 12 weeks
  Change in fasting plasma TG

SECONDARY OUTCOMES:
Area under the curve (AUC) for plasma TG | Baseline and the end of each 4 week treatment period for a total of 12 weeks
  Change in the total AUC for plasma TG from 0 to 8 hours following a high fat meal challenge.
Maximal Concentration (Cmax) and time to Cmax (Tmax) | Baseline and at the end of each 4 week treatment period for a total to 12 weeks
  Change in Cmax and Tmax for plasma TG for up to 8 hours following a high fat meal challenge.
Plasma TG during the OFTT | Baseline and at the end of each 4 week treatment period for a total of 12 weeks
  Change in plasma TG at 2, 4, 6, and 8 hours following a high fat meal challenge.
Fasting lipoprotein lipids | Baseline and at the end of each 4 week treatment period for a total of 12 weeks
  Change in fasting lipoprotein lipids, including high-density lipoprotein cholesterol (HDL-C), non-HDL-C, low-density lipoprotein cholesterol (LDL-C), and total cholesterol (TC).
Body weight | Baseline and at the end of each 4 week treatment period for a total of 12 weeks
  Change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lawson, MD, Principal Investigator — Biofortis; 211 East Lake Street; Addison, IL 60101
Locations (1):
- Biofortis, Addison, Illinois, United States

REFERENCES:
- [Background] Ables GP, Yang KJ, Vogel S, Hernandez-Ono A, Yu S, Yuen JJ, Birtles S, Buckett LK, Turnbull AV, Goldberg IJ, Blaner WS, Huang LS, Ginsberg HN. Intestinal DGAT1 deficiency reduces postprandial triglyceride and retinyl ester excursions by inhibiting chylomicron secretion and delaying gastric emptying. J Lipid Res. 2012 Nov;53(11):2364-79. doi: 10.1194/jlr.M029041. Epub 2012 Aug 21. PMID 22911105
- [Background] Cheng D, Iqbal J, Devenny J, Chu CH, Chen L, Dong J, Seethala R, Keim WJ, Azzara AV, Lawrence RM, Pelleymounter MA, Hussain MM. Acylation of acylglycerols by acyl coenzyme A:diacylglycerol acyltransferase 1 (DGAT1). Functional importance of DGAT1 in the intestinal fat absorption. J Biol Chem. 2008 Oct 31;283(44):29802-11. doi: 10.1074/jbc.M800494200. Epub 2008 Sep 3. PMID 18768481
- [Background] Chun OK, Chung SJ, Song WO. Estimated dietary flavonoid intake and major food sources of U.S. adults. J Nutr. 2007 May;137(5):1244-52. doi: 10.1093/jn/137.5.1244. PMID 17449588
- [Background] Denison H, Nilsson C, Kujacic M, Lofgren L, Karlsson C, Knutsson M, Eriksson JW. Proof of mechanism for the DGAT1 inhibitor AZD7687: results from a first-time-in-human single-dose study. Diabetes Obes Metab. 2013 Feb;15(2):136-43. doi: 10.1111/dom.12002. Epub 2012 Sep 30. PMID 22950654
- [Background] Martin SS, Blaha MJ, Elshazly MB, Toth PP, Kwiterovich PO, Blumenthal RS, Jones SR. Comparison of a novel method vs the Friedewald equation for estimating low-density lipoprotein cholesterol levels from the standard lipid profile. JAMA. 2013 Nov 20;310(19):2061-8. doi: 10.1001/jama.2013.280532. PMID 24240933
- [Background] Swinburn BA, Sacks G, Hall KD, McPherson K, Finegood DT, Moodie ML, Gortmaker SL. The global obesity pandemic: shaped by global drivers and local environments. Lancet. 2011 Aug 27;378(9793):804-14. doi: 10.1016/S0140-6736(11)60813-1. PMID 21872749
- [Background] Yen CL, Stone SJ, Koliwad S, Harris C, Farese RV Jr. Thematic review series: glycerolipids. DGAT enzymes and triacylglycerol biosynthesis. J Lipid Res. 2008 Nov;49(11):2283-301. doi: 10.1194/jlr.R800018-JLR200. Epub 2008 Aug 29. PMID 18757836